CLINICAL TRIAL: NCT04861311
Title: Testing the Efficacy of a Mindfulness- and Acceptance-Based Smartphone App Intervention for College Student Veterans With Posttraumatic Stress Disorder (PTSD): A Randomized Controlled Trial
Brief Title: Testing the Efficacy of a Mindfulness- and Acceptance-Based Smartphone App for PTSD: A Randomized Controlled Trial
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Principal Investigator, Andrew Thomas Reyes, Assistant Professor, University of Nevada, Las Vegas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1603895-3
Record Dates: First submitted 2021-04-22; First posted 2021-04-27 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Posttraumatic Stress Disorder, mindfulness, acceptance, resilience
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Mindfulness; Methods

STUDY DESIGN:
Intervention Model Description: Mindfulness/Acceptance-Based Smartphone App (MABSA) Intervention Group will use the smartphone app which comprises of audio-guided mindfulness meditations and video lessons. Participants are asked to listen to at least one guided meditation daily and watch one video lesson each week. Participants will also receive a weekly phone call for emotional and technical support. The wait-list control group will have the option to use the app-based intervention after 10 weeks of being in the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness/Acceptance-Based Smartphone App (MABSA) Intervention Group (Experimental): The intervention is 6 weeks in duration. Participants will be asked to listen daily to at least one audio-guided mindfulness meditation embedded in the app. They will also be asked to watch a weekly video lesson on mindfulness and acceptance and will be asked to write a reflection about the video. They will also receive weekly emotional and technical support during the duration of the intervention.
  Interventions: Behavioral: Mindfulness/Acceptance-Based Smartphone App (MABSA) Intervention
- Wait-List Control Group (No Intervention): The control group is a wait-list control group. Participants in the control group will be offered to use the app after 10 weeks of being in the study. The control group participants once they opted to use the app after 10 weeks will only have access to the app for 6 weeks.

INTERVENTIONS:
Behavioral: Mindfulness/Acceptance-Based Smartphone App (MABSA) Intervention — The intervention is based on the principles of Acceptance and Commitment Therapy (ACT). Therefore, the intervention is an ACT-based smartphone app delivered for 6 weeks in which participants will be applying the mindfulness and acceptance exercises embedded in the app. The mindfulness and acceptance exercises are audio-guided mindfulness meditations and video lessons about ACT.
  Arms: Mindfulness/Acceptance-Based Smartphone App (MABSA) Intervention Group

SUMMARY:
The purpose of the study is to test the feasibility and acceptability of a mindfulness- and acceptance-based smartphone app (MABSA) intervention for college student veterans with posttraumatic stress disorder (PTSD) symptoms. The study will use a randomized controlled trial design of two groups: intervention group of about 30 participants with PTSD and wait-list control group of about 30 participants. The duration of the MABSA intervention is 6 weeks. The following are the outcomes to be measured: resilience, PTSD, mindfulness, experiential avoidance, and rumination.

DETAILED DESCRIPTION:
The objective of the proposed study is to evaluate the feasibility of the Mindfulness/Acceptance-Based Smartphone App (MABSA) intervention in a randomized controlled trial (RCT) environment and to obtain generalized information (i.e., initial efficacy, recruitment, retention, adherence, satisfaction, and usability of the refined intervention). The expected results will provide the foundation for a prospective, fully powered, larger-scale RCT study. We previously developed the MABSA and pilot tested it in a single-arm study. Our central hypothesis is that the refined MABSA intervention would improve intervention satisfaction, app usability, and adherence and positively affect resilience, PTSD, mindfulness, experiential avoidance, and rumination. The specific aims of the proposed study are outlined below.

AIM 1: To refine the previously developed MABSA intervention. The 6-week smartphone-delivered program will involve (1) daily audio-guided meditations on various mindfulness and acceptance exercises constructed based on the principles of acceptance and commitment therapy; (2) weekly support and feedback through phone calls and/or texting the intervention facilitators; and (3) ecological momentary assessment (daily monitoring of PTSD and resilience) to monitor the progression of treatment response (i.e., the trajectory of resilience and PTSD recovery). We will obtain qualitative feedback on program content and format through a pilot test of the prototype with a group of eligible college student veterans (N = 4). Upon revising the intervention based on participants' feedback, we will develop the intervention protocol manual for the RCT.

AIM 2: To test the feasibility and acceptability of the refined MABSA intervention in a small-scale RCT for a prospective, fully powered, larger-scale RCT study. The small-scale RCT study will involve the following two groups of college student veterans: (1) the MABSA intervention group (N = 30) and the waitlist control group (N = 30). Upon collecting the data on recruitment, retention, adherence, intervention satisfaction, and app usability, we will determine the preliminary efficacy based on the following five outcomes: resilience, PTSD, mindfulness, experiential avoidance, and rumination. Qualitative feedback on the facilitators of and challenges to recruitment, retention, and adherence will be collected via exit interviews.

ELIGIBILITY:
Inclusion Criteria:

* (1) aged 18 years old or older, (2) currently registered as an undergraduate or graduate student, (3) has previous active military service from any U.S. military service branch, (4) has at least daily access to their own Apple iPhone (version 5 or later) or Android phone, and (5) have posttraumatic stress disorder (PTSD) symptoms (must have a score of 33 or above on the PTSD Checklist for DSM-5)

Exclusion Criteria:

* (1) Those who have a score of 32 or below on the PTSD Checklist for DSM-5 and (2) Those who have a cognitive impairment such as dementia-related disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
PTSD | We will measure PTSD at baseline, mid-intervention (Week 3), post-intervention (Week 6), and at one-month follow-up
  Changes in posttraumatic stress disorder (PTSD) symptoms based on the PTSD Checklist for DSM-5 (PCL-5)
Resilience | We will measure PTSD at baseline, mid-intervention (Week 3), post-intervention (Week 6), and at one-month follow-up
  Changes in resilience based on the Connor-Davidson Resilience Scale 25
Mindfulness | We will measure PTSD at baseline, mid-intervention (Week 3), post-intervention (Week 6), and at one-month follow-up
  Changes in mindfulness based on the Mindfulness Attention and Awareness Scale
Experiential Avoidance | We will measure PTSD at baseline, mid-intervention (Week 3), post-intervention (Week 6), and at one-month follow-up
  Changes in experiential avoidance based on the Acceptance and Action Questionnaire
Rumination | We will measure PTSD at baseline, mid-intervention (Week 3), post-intervention (Week 6), and at one-month follow-up
  Changes in rumination based on the Rumination Scale

SECONDARY OUTCOMES:
PTSD Recovery | We will measure PTSD daily using the app (ecological momentary assessment)
  Daily measures of PTSD using the abbreviated PTSD Checklist for DSM-5
Resilience Progression | We will measure resilience daily using the app (ecological momentary assessment)
  Daily measures of resilience using the abbreviate Connor-Davidson Resilience Scale 10

OTHER OUTCOMES:
Intervention Satisfaction | We will measure intervention satisfaction at mid-intervention (Week 3) and post-intervention (Week 6)
  Satisfaction with the intervention particularly on the areas of: overall satisfaction, perceived helpfulness, comprehension, intentions to use, and perceived fit
System Usability | We will measure perceived usability of the app at mid-intervention (Week 3) and post-intervention (Week 6)
  Perceived usability of the app using the System Usability Scale

CONTACTS AND LOCATIONS:
Overall Officials: Andrew T Reyes, PhD, Principal Investigator — University of Nevada, Las Vegas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reyes AT, Bhatta TR, Muthukumar V, Gangozo WJ. Testing the acceptability and initial efficacy of a smartphone-app mindfulness intervention for college student veterans with PTSD. Arch Psychiatr Nurs. 2020 Apr;34(2):58-66. doi: 10.1016/j.apnu.2020.02.004. Epub 2020 Feb 18. PMID 32248935
- [Background] Reyes AT, Serafica R, Sojobi A. College student veterans' experience with a mindfulness- and acceptance-based mobile app intervention for PTSD: A qualitative study. Arch Psychiatr Nurs. 2020 Dec;34(6):497-506. doi: 10.1016/j.apnu.2020.09.005. Epub 2020 Sep 11. PMID 33280672